CLINICAL TRIAL: NCT03541421
Title: Self-administration of Patients Own Drugs During Hospital Stay - Patient Involvement, Medication Errors and Health Economics
Brief Title: Self-administration of Patients Own Drugs During Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other); Hospital Pharmacy Central Denmark Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SAMRR2016_2019
Record Dates: First submitted 2017-10-25; First posted 2018-05-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-12

CONDITIONS: Patient Involvement; Medication Errors; Self Administration; Medication Adherence; Patient Satisfaction; Health Economics
MeSH Terms: conditions — Patient Participation; Medication Adherence; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The patients administers own drugs during hospital stay.
  Interventions: Other: Patient involvement in administration of drugs
- Control (No Intervention): The patients receive medications from the medicine room dispensed by a nurse (standard care). No intervention

INTERVENTIONS:
Other: Patient involvement in administration of drugs — The patient´s own drugs and an updated medication list will be placed in a lockable bedside table. During hospitalization the patient is responsible for taking his own medication. If a new drug is prescribed, the patient will be involved and instructed about it. Furthermore the smallest package will be delivered so that the patient can begin self-administration of the new drug during hospitalization.
  Arms: Intervention

SUMMARY:
Background Medication administration errors occur in around 20% of administrations. Patient involvement (PI) is recommended and self-management support e.g. as self-administration of patient's own drugs during hospital stay is a central component of practising PI.

Aim To investigate whether PI in administering drugs in hospital affects the number of medication errors, medication adherence and patient satisfaction and whether it is economically advantageously.

Materials and methods The PhD Study is performed at the Department of Cardiology, Randers Regional Hospital.

The study design is "complex intervention" and the PhD study therefore consists of three studies. In study 1 the intervention is developed, investigated for feasibility and pilot-tested in small scale. In study 2 and 3 the intervention is evaluated within a RCT with outcomes as medication errors, medication adherence, patient satisfaction and cost-effectiveness.

DETAILED DESCRIPTION:
Background When patients are admitted to Danish hospitals, the responsibility for their medication is taken over by the hospital staff.

Medication administration errors occur in approximately 20% of the total opportunities for error.

Patient involvement (PI) is recommended and self-management support is a central component of PI aiming to improve patients' knowledge, skills and confidence into managing their health condition. "Self-administration of patient's own drugs" during hospital stay is considered a central part of self-management support.

Self-administration of patient's own drugs has been tested in the Capital Region of Denmark. Conclusions were that self-administration increase PI, prepare patients to manage their medication after discharge and release resources within the care group. The occurrence of medication errors compared to traditional medication system was not investigated.

Aim The aim is to investigate whether PI in administering drugs during hospital stay affects the number of medication errors, medication adherence and patient satisfaction and whether it is economically advantageously.

Materials and methods The study design is "complex intervention" and a stepwise process is recommended by the UK Medical Research Council. In study 1 the intervention will therefore be developed, investigated for feasibility and pilot-tested in small scale. In study 2 and 3 the intervention will be evaluated within a RCT.

Intervention If the patient is assessed able to self-administer own drugs at admission, the patient will be asked if he has brought (or can get someone to bring) his usual drugs to hospital. The drugs and an updated medication list will be placed in a lockable bedside table. During hospitalization the patient is responsible for taking his own medication. If a new drug is prescribed, the patient will be involved and instructed about it. Furthermore the smallest package will be delivered so that the patient can begin self-administration of the new drug during hospitalization. After discharge, the patient can bring the package and an updated medication list back home to ensure continuity in the medical treatment.

Study 1: Feasibility and pilot study The PhD study is performed at the Department of Cardiology, Randers Regional Hospital. By visits in the department it is assessed how many eligible patients there are, how many patients change ability to self-administer own drugs during hospital stay (risk of withdrawal), how many drugs do they receive and how many opportunities for error are there? These numbers will be used to assess the inclusion period and to calculate the sample size for the RCT. The intervention and workflows will be developed in collaboration with nurses, physicians and patients to ensure acceptability, feasibility and high patient safety.

In the pilot study the intervention and tools for study 2 is tested.

Study 2: RCT The study is a randomized controlled trial where patients are randomized for either intervention or control. The intervention group consists of patients who self-administer own drugs at home and are able to self-administer own drugs during hospital stay. The control group consists of patients who self-administer own drugs at home, who is able to self-administer own drugs during hospital stay, but where standard care is used (not self-administration).

Study 3: Health economic evaluation The cost effectiveness of the intervention is assessed from the perspectives of the hospital and the health system. Relevant resource use will be identified and detailed in study 1 and measured alongside the RCT.

The costs incurred in the intervention group will be compared to the control group based on an intention to treat principle. If the intervention costs in the intervention group exceed those in the control group, the costs will be related to an effect measure such as number of medication errors avoided.

Perspectives When the patient plays an active role in their own medication, it is expected that they will have a more comprehensive and adequate understanding of their situation and will be better to manage their own medication. The number of medication errors during the processes of dispensing and administering drugs at the wards is expected to decrease when patients administers their own drugs. PI and the use of patient's own drugs during admission are expected to contribute to a better utilization of the resources of the Health Care System.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the department "Medicinsk sengeafsnit 1", at Randers Regional Hospital Monday to Friday from 8.00 am to 6.00 pm
* Patients who are self-administering own drugs at home

Exclusion Criteria:

* Patients under 18 years old
* Patients who are not able to self-administer own drugs during hospital stay
* Patients who do not speak Danish
* Patients who can not or will not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Medication administration errors | on the day of inclusion and the following day. 1-2 days.
  The total number of medication administration errors observed compared to the total opportunities for error. Direct observation of nurses (control group) and patients (intervention group) dispensing drugs.

SECONDARY OUTCOMES:
Medication errors after discharge | 14 days after discharge
  Discrepancies in medicationlists 14 days after discharge through interviews
Medication Adherence | at hospitalization and 14 days after discharge
  The patients medication adherence is assessed through interviews
Patient satisfaction | 14 days after discharge
  The patients satisfaction with the hospital stay is assessed through interviews
Health economics | from day of inclusion to day of discharge (1-31 days).
  The cost effectiveness of the intervention is assessed. The costs incurred in the intervention group will be compared to the control group based on an intention to treat principle. If the intervention costs in the intervention group exceed those in the control group, the costs will be related to an effect measure such as number of medication errors avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte A. Sørensen, Ph.d.student, Principal Investigator — Health, Aarhus University
Locations (1):
- Medicinsk Sengeafsnit 1, Regionshospitalet Randers, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen CA, Olesen C, Lisby M, Enemark U, de Thurah A. Self-administration of medication during hospitalization-a randomized pilot study. Pilot Feasibility Stud. 2020 Aug 18;6:116. doi: 10.1186/s40814-020-00665-3. eCollection 2020. PMID 32821422